CLINICAL TRIAL: NCT02052427
Title: Adipose-derived Regenerative Cells in the Treatment of Patients With Chronic Ischemic Heart Disease Not Amenable to Surgical or Interventional Revascularization II
Brief Title: Safety & Efficacy of Adipose-Derived Regenerative Cells in the Treatment of Chronic Myocardial Ischemia (ATHENA II)
Acronym: ATHENA II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cytori Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATHENA II
Record Dates: First submitted 2014-01-30; First posted 2014-02-03 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Myocardial Ischemia
Keywords: Ischemic heart disease; Coronary artery disease; Chronic Heart Failure; Cardiovascular disease; adult stem cells; adipose derived regenerative cells
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ADRCs (Experimental): Adipose-Derived Regenerative Cells (ADRCs) processed by the Celution System:
  * 0.8 x 10^6 cells/kg body weight (not to exceed 80.0 x 10^6 cells)
  * Delivered via the MYOSTAR™ Injection Catheter in 15 intramyocardial injections
  Interventions: Device: Celution System
- Placebo (Placebo Comparator): Placebo - Physiological Solution
  * Inactive substance (Lactated Ringers + autologous blood)
  * Delivered via the MYOSTAR™ Injection Catheter in 15 intramyocardial injections
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Celution System — ADRCs processed by the Celution System for reintroduction into the myocardium
  Arms: ADRCs
Device: Placebo — Physiological solution made of Lactated Ringers solution and a small amount (<1mL) of autologous blood
  Arms: Placebo

SUMMARY:
This is a prospective, randomized, placebo-controlled, double blind safety and efficacy clinical trial.

DETAILED DESCRIPTION:
To assess the safety and efficacy of Adipose-Derived Regenerative Cells (ADRCs) delivered via an intramyocardial route in the treatment of chronic ischemic heart disease in patients who are not eligible for percutaneous or surgical revascularization.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females > 20 and < 80 years of age
2. Significant multi-vessel coronary artery disease not amenable to percutaneous or surgical revascularization
3. CCS Angina Functional Class II-IV and/or NYHA Stages of Heart Failure Class II or III
4. On maximal medical therapy for anginal symptoms and/or heart failure symptoms
5. Hemodynamic stability (SBP ≥ 90 mm/Hg, HR <110)
6. Ejection fraction ≥ 20% and ≤ 45%
7. Inducible ischemia using an objective assessment of ischemia within 1 year of screening (i.e. exercise ECG changes, SPECT)
8. Left ventricular wall thickness ≥ 8 mm at the target site for cell injection

Exclusion Criteria:

1. Atrial fibrillation or flutter without a pace maker that guarantees a stable heart rate
2. Unstable angina
3. LV thrombus, as documented by echocardiography
4. Planned staged treatment of CAD or other intervention on the heart
5. Platelet count < 100,000/mm3
6. WBC < 2,000/mm3
7. TIA or stroke within 90 days prior to randomization
8. ICD shock within 30 days prior to randomization
9. Any condition requiring immunosuppressive medication
10. A high-risk acute coronary syndrome (ACS) or a myocardial infarction in the 60 days prior to randomization
11. Revascularization within 60 days prior to randomization
12. Inability to walk on a treadmill except for class IV angina patients who will be evaluated separately
13. Hepatic dysfunction, as defined as aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 1.5 times the upper limit of normal range (x ULN)
14. Hemoglobin ≤ 10.0 g/dL

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-01; Primary Completion 2015-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy - Change in Minnesota Living with Heart Failure Questionnaire | 6 months post treatment
  Change in Minnesota Living with Heart Failure Questionnaire prior to treatment and at 6 months post treatment.

SECONDARY OUTCOMES:
Secondary Efficacy - Change in mVO2 | 6 months post treatment
  Change in mVO2 at 6 months as assessed by Exercise Tolerance Test
Secondary Efficacy - Change in LVESV/LVEDV | 6 months post treatment
  Change in LVESV/LVEDV at 6 months as assessed by Echocardiography
Secondary Efficacy - Change in Ejection Fraction | 6 months post treatment
  Change in Ejection Fraction (%) at 6 months assessed by 2D Contrast Echocardiography
Secondary Efficacy - Change in perfusion defect | 6 months post treatment
  Change in perfusion defect at 6 months assessed by Rest/Pharmacologic Stress SPECT
Secondary Efficacy - Resource Utilization | through 12 months post treatment
  Resource utilization - hospital length of stay, re-hospitalization for cardiac related events
Secondary Efficacy - Change in heart failure symptoms, angina, and quality of life | through 12 months post treatment
  Change in heart failure symptoms, angina, and quality of life assessed by - NYHA classification, CCS classification, MLHFQ (other than 6 months)

OTHER OUTCOMES:
Safety - Number of Patients Experiencing Treatment Emergent SAEs | Treatment through 12 months
Safety - Number of Patients Experiencing Arrhythmias Assessed via Holter monitor | Screening through 3 months post treatment
Safety - Number of patients that experience a MACE | Treatment through 12 months
  Number of patients that experience a Major Adverse Cardiac Event (MACE)

CONTACTS AND LOCATIONS:
Overall Officials: Emerson C. Perin, MD, PhD, Principal Investigator — The Stem Cell Center at Texas Heart Institute; Timothy Henry, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- University Hospital Case Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Result] Henry TD, Pepine CJ, Lambert CR, Traverse JH, Schatz R, Costa M, Povsic TJ, David Anderson R, Willerson JT, Kesten S, Perin EC. The Athena trials: Autologous adipose-derived regenerative cells for refractory chronic myocardial ischemia with left ventricular dysfunction. Catheter Cardiovasc Interv. 2017 Feb 1;89(2):169-177. doi: 10.1002/ccd.26601. Epub 2016 Sep 23. PMID 27148802